CLINICAL TRIAL: NCT00379028
Title: A Randomized, Double-blind, Two-way Cross-over Study Evaluating Systemic Bioavailability and Airway Clearance of SymbicortTurbuhaler 320/9mcg vs SeretideDiskus 50/500mcg After Single Inhalations in Patients With COPD and Healthy Volunteers
Brief Title: Airway Clearance Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D5892C00012; EUDRACT 2006-002412-10
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: Budesonide/Formoterol Turbuhaler
  Other Names: Symbicort
Drug: Salmeterol/Fluticasone Diskus

SUMMARY:
The purpose of the study is to evaluate how the airways in COPD patients, compared to healthy volunteers, absorb steroid drugs from Symbicort Turbuhaler and Seretide Diskus. The blood concentrations of the steroids will be used as surrogate marker.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients: ≥40 years of age, Diagnosed COPD with symptoms ≥1 year, Pre-bronchodilatory FEV1 ≤55% of PN, Productive cough with expectoration.
* Healthy volunteers: ≥18 years of age, Healthy, Pre-bronchodilatory FEV1 >80% of PN, Non-smoker

Exclusion Criteria:

* COPD patients: Current respiratory tract disorder other than COPD, Asthma before 40 years of age, Significant or unstable cardiovascular disorder,
* Healthy volunteers: Use of any regular medication or therapy, Pregnancy or breast-feeding,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-09; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of the plasma concentrations of the steroid components 0 - 10 hours after study drug inhalation in patients with COPD and healthy volunteers

SECONDARY OUTCOMES:
Exploratory investigations on the amount of steroids expectorated spontaneously in COPD patients
Correlation between baseline lung function and AUC of steroids after inhalation.

CONTACTS AND LOCATIONS:
Overall Officials: Christer Hultquist, MD, Study Director — AstraZeneca; Tim Harrisson, MD, Principal Investigator — Nottingham University
Locations (2):
- Research Site, Lund, Sweden
- Research Site, Nottingham, United Kingdom

REFERENCES:
- [Derived] Dalby C, Polanowski T, Larsson T, Borgstrom L, Edsbacker S, Harrison TW. The bioavailability and airway clearance of the steroid component of budesonide/formoterol and salmeterol/fluticasone after inhaled administration in patients with COPD and healthy subjects: a randomized controlled trial. Respir Res. 2009 Oct 31;10(1):104. doi: 10.1186/1465-9921-10-104. PMID 19878590